CLINICAL TRIAL: NCT03629821
Title: Effect of Classic Ballet Practice on School Children's Postural Balance: Randomized Clinical Trial
Brief Title: Effect of Classic Ballet Practice on School Children's Postural Balance
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: The study has been suspended because COVID pandemic.
Sponsor: Universidade Federal de Santa Maria (Other)
Responsible Party: Principal Investigator, Karine Josibel Velasques Stoelben, Principal Investigator, Universidade Federal do Pampa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 65327017.2.0000.5346
Record Dates: First submitted 2018-06-11; First posted 2018-08-14 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Child, Only
Keywords: Postural Balance; Dance Therapy; Exercise Therapy

STUDY DESIGN:
Intervention Model Description: Two groups design where one group receives treatment and the other not in the same period of time.
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ballet (Experimental): Subjects who will receive the experimental protocol.
  Interventions: Other: Ballet
- Control (No Intervention): Subjects who will not receive the experimental protocol, only will be on a wait list.

INTERVENTIONS:
Other: Ballet — The classic ballet classes will respect biological limits of children. The sessions will be 75 minutes long, twice a week during 8 weeks. The class sequence will be: warm-up, follow by exercises about upper and lower limbs ballet positions and sequences of ballet jumps, and at the end a cool-down.
  Arms: Ballet

SUMMARY:
Is a parallel longitudinal protocol where half patients receive a experimental protocol and the other half receive orientation to maintain your daily live routine as usually. The experimental protocol include Ballet sessions. The hypothesis is interventional group will improve the balance control more than control group.

ELIGIBILITY:
Inclusion Criteria:

* Female sex
* 9 to 12 years of age

Exclusion Criteria:

* Musculoskeletal pain at last 3 months
* Perform other physical activity besides scholar's physical activity
* Has been participated Ballet class.

Ages: 9 Years to 12 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2018-07-15 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in total score of Star Excursion Balance Test at 8 weeks. | Before, immediate after intervention protocol
  Changing between the beginning and end of intervention. This measure is shown in cm.
Change from baseline in anteriorposterior and mediolateral displacements of Pressure Center at 8 weeks. | Before, immediate after intervention protocol
  Changing between the beginning and end of intervention of anteroposterior and mediolateral displacements of pressure center in cm.
Change from baseline in average speed of Pressure Center at 8 weeks. | Before, immediate after intervention protocol
  Changing between the beginning and end of average speed of pressure center in cm/s.
Change from baseline in 95% ellipse area of Pressure Center at 8 weeks. | Before, immediate after intervention protocol
  Changing between the beginning and end of 95% ellipse area of pressure center in cm².
Maintenance at 30 and 60 days from baseline in total score of Star Excursion Balance Test. | Immediate after, 30 and 60 days after intervention protocol.
  Changing between the end and 30 and 60 days after intervention. This measure is shown in cm.
Maintenance at 30 and 60 days from baseline in anteroposterior and mediolateral displacements of pressure center | Immediate after, 30 and 60 days after intervention protocol.
  Changing between the end and 30 and 60 days after intervention of anteroposterior and mediolateral displacements of pressure center in cm.
Maintenance at 30 and 60 days from baseline in average speed of pressure center | Immediate after, 30 and 60 days after intervention protocol.
  Changing between the end and 30 and 60 days after intervention of average speed of pressure center in cm/s.
Maintenance at 30 and 60 days from baseline in 95% ellipse area of pressure center | Immediate after, 30 and 60 days after intervention protocol.
  Changing between the end and 30 and 60 days after intervention of 95% ellipse area of pressure center in cm².

SECONDARY OUTCOMES:
Vertical stiffness | Before, immediate after, 30 and 60 days after intervention protocol
  Stiffness estimate by force plate data and displament of center of mass
Peak and absortion rate of ground reaction force | Before, immediate after, 30 and 60 days after intervention protocol
  Greatest value and absortion rate (between inicial contat and peak) of ground reaction force

OTHER OUTCOMES:
Physical activity level | Before intervention
  Assessed by final score of Physical Activity Questionnaire for Children. The score questions are about daily physical activity of children. Final score is a mean calculate by 9 items/questions with range 1 to 5. A final score of 1 (minimum) indicates low physical activity, whereas a score of 5 (maximum) indicates high physical activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Kelen Munhos Pinto, Santa Maria, Rio Grande do Sul, Brazil